CLINICAL TRIAL: NCT03227549
Title: Investigating the Direct Superior Approach for Total Hip Arthroplasty as an Effective Alternative to Traditional Posterior Approach
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: THA DSA
Record Dates: First submitted 2017-06-22; First posted 2017-07-24 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Total Hip Arthroplasty
MeSH Terms: interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Direct Superior Approach (Experimental): The intervention being tested is the surgical approach.
  Interventions: Procedure: Direct Superior Approach; Device: Total Hip Arthroplasty
- Posterior Approach (Active Comparator)
  Interventions: Device: Total Hip Arthroplasty; Procedure: Posterior Approach

INTERVENTIONS:
Procedure: Direct Superior Approach — Total hip arthroplasty using direct superior approach
  Arms: Direct Superior Approach
Device: Total Hip Arthroplasty — Total Hip Arthroplasty using direct superior or posterior approach
Procedure: Posterior Approach — Total Hip Arthroplasty using posterior approach
  Arms: Posterior Approach

SUMMARY:
Hip replacement surgery is an effective option for treating pain and functional impairment in chronic hip conditions. Various surgical approaches have been developed to expose the hip joint for the procedure, each with advantages and disadvantages. The posterior approach (PA) to total hip replacement is a commonly used exposure method. This approach involves a large incision and requires multiple cuts through muscle and other soft tissues to expose the hip joint. Despite excellent outcomes, the PA is known to have an increased rate of dislocation compared to other exposures. The direct superior (DS) approach has been developed to improve the PA by decreasing the amount of soft tissue injury at the time of surgery and improving postoperative stability. The DS approach involves a much shorter incision and reduces the need to damage as much soft tissues surrounding the hip joint during exposure. Specialized equipment developed for this technique allows the surgeon to place the hip replacement components. The proposed research study is designed to address a deficit in knowledge regarding outcomes on patients who have had a DS approach for total hip arthroplasty. This study will provide much needed insight into the advantages and disadvantages of the DS approach as compared to PA for total hip arthroplasty.

DETAILED DESCRIPTION:
The primary objective of this study is to compare the health status and functional outcomes of patients who have undergone total hip arthroplasty (THA) utilizing the direct superior (DS) approach to those who have undergone THA utilizing the posterior approach (PA). The aim is to quantify changes in functional status using accelerometer-based gait analysis and self-reported questionnaires, and to assess peri-operative recovery including narcotic use, length of stay, blood loss, complications and readmission for any reason.

It is hypothesized that patients who undergo THA utilizing the DS approach will have more favorable results in terms of health status and functional outcomes when compared to those who receive the PA approach. It is expected that patients in the DS group will display an earlier improvement in gait postoperatively, will have a shorter length of stay in hospital, and will have decreased postoperative pain as measured by narcotic use. No measurable difference in the position of the THA implants is expected between groups.

The proposed clinical study is a prospective randomized trial of 80 patients undergoing total hip arthroplasty utilizing either a PA or DS approach. Postoperative outcomes including narcotic use, length of stay and complications will be abstracted from the chart and any readmissions will be documented. Follow-up exams will occur at 6 weeks, 6 months, 12 months and 24 months from time of surgery. Radiographic evaluation will be performed at each interval to assess the position of the implants. Gait symmetry data will be collected pre-operatively as well as at 6 months, 12 months, and 24 months and will be assessed for longitudinal changes in characteristics such as stride frequency, envelope, surge, lurch and functional leg length discrepancy. Health status, functional outcome, and patient quality of life measures will be recorded at all follow-up intervals. Joint function will be assessed before and after surgery using the EuroQol questionnaire, Oxford 12 Hip questionnaire, Self-Administered Comorbidity Questionnaire (SCQ), visual analogue scales (VAS) for pain and satisfaction, and UCLA Activity Level Scale. Rates of infection, instability and revision for any cause will be monitored for the duration of the 2 year follow-up.

Pre-operative subject characteristics will be compared between groups using Student's t-tests (unpaired, two-sided). For the post-operative follow-up questionnaire and radiographic data, two-way repeated measures analyses of variance (ANOVA) for group differences will be used to analyze data collected at multiple time points. Gait data will be analyzed using Gaitview software.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic osteoarthritis of the hip indicating surgical intervention
* Uncemented femoral stem and acetabular cup indicated
* Patients between the ages of 18 and 80, inclusive.
* Ability to give informed consent

Exclusion Criteria:

* Patients less than 18 years of age, or 81 years of age and older
* Active or prior infection of the affected hip
* Morbid obesity (BMI > 45)
* Medical condition precluding major surgery
* Severe osteoporosis or osteopenia
* Neuromuscular impairment
* Patients with known or tested-positive allergy to metals
* Pregnancy

Ages: 18 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2025-07-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
EQ-5D patient reported outcome measure | 2 years
  Health status measure
Oxford-12 patient reported outcome measure | 2 years
  Functional outcome measure

SECONDARY OUTCOMES:
Length of stay | 0 - 30 days
  Time until discharge from hospital following surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Capital District Health Authority, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No